CLINICAL TRIAL: NCT01627548
Title: UCLA Welcome Back Veterans Family Resilience Center Couples Counseling for Combat Veterans
Brief Title: UCLA Couples Counseling for Combat Veterans
Acronym: CCCV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Proposed studies were not funded
Sponsor: University of California, Los Angeles (Other)
Collaborators: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shirley Glynn, Associate Researcher, University of California, Los Angeles
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 11-003109
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: PTSD; Recent Era Combat Veteran; Couples Communication
Keywords: PTSD; Couples; Combat Veteran; Warfighter; OEF; OIF; OND; Structured Approach Therapy; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlisted Intervention (Active Comparator): Couple will be consented, assessed and randomized to a waitlist of 4 months. The couple will be reassessed at 8 weeks and prior to initiating intervention.
  Interventions: Behavioral: Structured Approach Therapy
- Immediate Intervention (Active Comparator): Eligible couples who are randomized to immediate intervention will begin sessions with a trained interventionist within weeks of consent and initial assessments
  Interventions: Behavioral: Structured Approach Therapy

INTERVENTIONS:
Behavioral: Structured Approach Therapy — The SAT treatment is provided in 12 weekly 50-minute sessions and is fully manualized. First, couple-based exposure techniques are used to address anxiety about intimacy, increasing the traumatized person's ability to engage in social and relational behaviors that promote bonding and satisfaction. Second, as anxiety decreases, couple-based techniques are also used to increase the positive experiences the couple is having. These activities expose the traumatized person to positive feelings instead of anxiety, so that he/she may become desensitized to the anxiety caused by the closeness, and more comfortable engaging in intimate behaviors.

SUMMARY:
A pilot intervention of an existing intervention adapted for the returning warfighter population: a couples treatment for PTSD, Structured Approach Therapy (SAT), which emphasizes reducing the PTSD avoidance/numbing symptoms that are corrosive in families.

ELIGIBILITY:
Inclusion Criteria:

* OIF/OEF/ OND veteran with at least one deployment
* In a cohabitating relationship for 6 months or longer
* Cohabitating 50% of the time or more
* Diagnosed with PTSD or meets the diagnosis criteria for PTSD as related to deployment experience (CAPS)
* Ability to make weekly appointments
* Willingness to commit to change

Exclusion Criteria:

* Receiving an evidence-based treatment for PTSD within the past 6 months
* Receiving couples therapy within the last 6 months
* Moderate or excessive physical violence within the past 3 months (CTS)
* Alcohol/substance dependence (SCID)
* Known domestic violence/abuse (CTS)
* Symptoms of psychosis within the past 3 months
* Unstable psychiatric medicine usage or on regimen less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Improved couples communication as measured by standardized assessments | 4-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shrley M Glynn, PhD, Principal Investigator — University of California, Los Angeles; Patricia E Lester, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States